CLINICAL TRIAL: NCT02967614
Title: A Randomized, Open-label, 2-period, Parallel Group, Multiple-dose Study to Evaluate the Drug-drugs Interaction Between Dorzolamide and Brimonidine in Healthy Korean Male Volunteers
Brief Title: KJ-TFC-004 Drug-drug Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kukje Pharma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KJ-TFC-004
Record Dates: First submitted 2016-11-12; First posted 2016-11-18 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2016-11

CONDITIONS: Glaucoma; Eye Diseases; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Eye Diseases; Ocular Hypertension | interventions — Brimonidine Tartrate, Timolol Maleate Drug Combination; dorzolamide; Brimonidine Tartrate; Timolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- [A]→[A]+[B] (Experimental): Period 1 : At each dosing of Treatment A eye drops is administered for 8days
  Period 2 : At each dosing of Treatment A + Treatment B eye drops is administered for 92days
  Interventions: Drug: [A]; Drug: [A]+[B](1)
- [B]→[A]+[B] (Experimental): Period 1 : At each dosing of Treatment B eye drops is administered for 92days
  Period 2 : At each dosing of Treatment A + Treatment B eye drops is administered for 8days
  Interventions: Drug: [B]; Drug: [A]+[B](2)

INTERVENTIONS:
Drug: [A] — One eye drop(about 40ul) / Day1 ~ Day8 / BID
  Other Names: Brimonidine , Timolol
  Arms: [A]→[A]+[B]
Drug: [B] — One eye drop(about 40ul) / Day1 ~ Day92 / BID
  Other Names: Dorzolamide
  Arms: [B]→[A]+[B]
Drug: [A]+[B](1) — One eye drop(about 40ul) / Day9 ~ Day100 / BID
  Other Names: Brimonidine , Timolol , Dorzolamide
  Arms: [A]→[A]+[B]
Drug: [A]+[B](2) — One eye drop(about 40ul) / Day93 ~ Day100 / BID
  Other Names: Brimonidine , Timolol , Dorzolamide
  Arms: [B]→[A]+[B]

SUMMARY:
To assess the pharmacokinetic Interaction between Dorzolamide and Brimonidine in healthy male subjects.

DETAILED DESCRIPTION:
Clinical trial to evaluate the influence of drug and drug-drug interactions of Brimonidine and Dorzolamide co-administration on the pharmacokinetics of Brimonidine and pharmacokinetics of Dorzolamide in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male adults aged between 19 and 50 during screening period
* BMI more than 18kg / m2 and less than 30kg / m2 and weight more than 55kg
* Signed the informed consent form prior to study participation.

Exclusion Criteria:

* Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in kidney, liver, cardiovascular system, respiratory system, endocrine system, or neuropsychiatric system.

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-12; Primary Completion 2017-12 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of Brimonidine and Dorzolamide | pre- and post dose of Brimonidine and Dorzolamide administration]
  Group 1 Brimonidine Period 1 : 1d 0h,7d 0h,7d 12h,8d 0h(pre-dose), 8d 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12 h post-dose (Total 15 Point)
  Period 2 : 9d 0h,23d 0h,37d 0h,51d 0h,65d 0h,79d 0h,93d 0h,99d 0h,99d 12h, 100d 0h(pre-dose),100d 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12 h post-dose (Total 21Point)
  Dorzolamide
  Period 2 : 9d 0h,23d 0h,37d 0h,51d 0h,65d 0h,79d 0h,93d 0h,99d 0h,99d 12h,100d 0h (pre-dose), 100d 0.25,0.5,0.75,1,1.5,2,2.5,3,4,8,12 h post-dose (Total 21Point)
  Group 2 Brimonidine Period 2 : 93d 0h,99d 0h,99d 12h,100d 0h(pre-dose),100d 0.25, 0.5, 0.75, 1, 1.5,2,2.5,3,4,8,12h post-dose (Total 15Point)
  Dorzolamide Period 1 : 1d 0h, 15d 0h, 29d 0h, 43d 0h, 57d 0h, 71d 0h, 85d 0h, 91d 0h, 91d 12h, 92d 0h (pre-dose), 92d 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12 h post-dose (Total 21Point)
  Period 2 : 93d 0h, 99d 0h, 99d 12h, 100d 0h (pre-dose), 100d 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12 h post-dose (Total 15Point)

SECONDARY OUTCOMES:
Trough concentration of Dorzolamide and N-Desethyl-Dorzloamide | pre- and post dose of Dorzolamide and Dorzloamide administration]
  Group 1 Brimonidine Period 1 : 1d 0h,7d 0h,7d 12h 8d 0h (pre-dose),8d 0.25,0.5,0.75,1,1.5,2,2.5,3, 4,8,12 h post-dose (Total 15Point)
  Period 2 : 9d 0h,23d 0h,37d 0h,51d 0h,65d 0h,79d 0h,93d 0h,99d 0h,99d 12h,100d 0h (pre-dose),100d 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12h post-dose (Total 21Point)
  Dorzolamide
  Period 2 : 9d 0h,23d 0h,37d 0h,51d 0h,65d 0h,79d 0h,93d 0h,99d 0h,99d 12h,100d 0h (pre-dose), 100d 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12h post-dose (Total 21Point)
  Group 2 Brimonidine Period 2 : 93d 0h,99d 0h,99d 12h,100d 0h (pre-dose),100d 0.25, 0.5, 0.75, 1, 1.5,2,2.5,3,4,8,12h post-dose (Total 15Point)
  Dorzolamide Period 1 : 1d 0h,15d 0h,29d 0h,43d 0h,57d 0h,71d 0h,85d 0h,91d 0h, 91d 12h,92d 0h(pre-dose), 92d 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12h post-dose (Total 21Point)
  Period 1 : 93d 0h,99d 0h,99d 12h,100d 0h (pre-dose), 100d 0.25, 0.5, 0.75, 1, 1.5,2,2.5,3,4,8,12h post-dose (Total 15Point)

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-sang Yu, Ph.d., M.B.A, Principal Investigator — Clinical Trial Center, Seoul National University Hospital
Locations (1):
- Clinical Trial Center, Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No